CLINICAL TRIAL: NCT02451696
Title: A Pilot Study To Evaluate The Effects of Everolimus on Brain mTOR Activity and Cortical Hyperexcitability in TSC and FCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-00245
Record Dates: First submitted 2014-10-08; First posted 2015-05-22 (Estimated); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy; Tuberous Sclerosis Complex; Focal Cortical Dysplasia
MeSH Terms: conditions — Epilepsy; Tuberous Sclerosis; Focal Cortical Dysplasia | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treated Subjects (Experimental): This group will be treated with everolimus 7-28 days prior to surgery
  Interventions: Drug: Everolimus
- Reference Subjects (No Intervention): This group will be enrolled as reference subjects, and will be undergoing routine surgery as part of standard of care treatment. No intervention will be provided to these subjects as part of the study.

INTERVENTIONS:
Drug: Everolimus — This study will measure if the drug called Everolimus effects mTOR signaling (an electrical activity signal in the brain) in patients with Tuberous Sclerosis Complex (TSC) and Focal Cortical Dysplasia (FCD) with treatment resistant epilepsy (TRE) who will be undergoing brain surgery. One group of patients will be treated with Everolimus, for 7-28 days prior to epilepsy surgery and another will not. We will determine if there is a difference in mTOR signaling between the patients who were treated with Everolimus and those who were not
  Other Names: Trade Name: Afinitor®
  Arms: Treated Subjects

SUMMARY:
The purpose of this study is to measure if the drug called Everolimus effects mTOR signaling (an electrical activity signal in the brain) in patients with Tuberous Sclerosis Complex (TSC) and Focal Cortical Dysplasia (FCD) with treatment resistant epilepsy (TRE) who will be undergoing brain surgery. One group of patients will be treated with Everolimus, and another will not. Researchers will determine if there is a difference in mTOR signaling between the patients who were treated with Everolimus and those who were not. Previous studies have suggested that Everolimus may reduce seizure activity in TSC patients by decreasing mTOR signaling. Since patients with FCD may also have excess mTOR signaling brain activity, Everolimus may also reduce seizure activity in these patients.

The drug Everolimus is approved by the Food and Drug Administration to treat specific types of breast, pancreatic, and kidney cancer, a kidney tumor called an angiomyolipoma (common in patients with TSC), and TSC patients who have a brain tumor called a subependymal giant cell astrocytoma (SEGA). However, in this research it is considered to be an investigational since it is not approved for reduction in mTOR signaling and a decrease in seizure frequency. Researchers believe that Everolimus may be useful in reducing something called cortical hyperexcitability, which is the excess brain activity that can contribute to seizures.

DETAILED DESCRIPTION:
This is a single center open-label pilot clinical trial of patients with TRE, ages 1 to 40 years old, with TSC or FCD who are scheduled for epilepsy surgery. Patients will be treated with everolimus for 7 to 28 days prior to epilepsy surgery with extension of time from 7 to 28 days in successive cohorts of patients. The initial cohort of at least three patients will be treated for 7 days and after the safety of therapy is assured for this group, there will be an extension of the treatment to 14 days for at least three patients. This will be extended at one week intervals/three patient groups to a maximum treatment duration of 28 days. Resected brain tissue will be analyzed for activation of mTORC1 and mTORC2 signaling pathways, glutamatergic and GABA-ergic neurotransmission using histochemistry, genetic analysis, as well as extracellular field recordings in acute ex-vivo brain slices from surgery. A blood sample, collected at the time of surgery, will be analyzed for everolimus levels and VEGF-D. All patients will undergo standardized intra-operative ECoG recordings over the primary epileptogenic region and reviewed blindly.

Subjects will be in the study for 7-28 days. The investigators will study variables listed in specific aims 1 and 2 in TSC and FCD patients treated with 7 to 28 days of everolimus and compare these to untreated control patients with TRE and TSC or FCD. A concurrent comparison group of 12 subjects will also be enrolled. They will all be undergoing routine surgery for the diagnosis of TRE with TSC or FCD.

All study procedures will be performed at the Comprehensive Epilepsy Center (CEC) with the exception of the surgery, which will be performed at Tisch Hospital.

ELIGIBILITY:
Inclusion Criteria

1. Patients: 1 year to 40 years. 2. Diagnosis: treatment resistant epilepsy due to Tuberous Sclerosis Complex or Focal Cortical Dysplasia Inclusion Criteria (Concurrent Comparison Group)

1. Patients: 1 year to 40 years. Matched for age (+/- 7 years) and sex of subjects in the treatment group.
2. Diagnosis: treatment resistant due to TSC or FCD. Matched for diagnosis of TSC and FCD.
3. Brain surgery for seizure control in which tissue is banked for research utilizing an existing IRB-approved study.

Exclusion Criteria

1. Treatment with an mTOR inhibitor (everolimus, sirolimus) during the past four weeks.
2. Known hypersensitivity to an mTOR inhibitor (everolimus, sirolimus)
3. Failure to establish diagnosis of treatment resistant epilepsy (i.e., adequate trials of two appropriately-chosen, tolerated and adequate trials of antiepileptic drugs) [32].
4. Exposure to any investigational agent in the month prior to study entry.
5. History of malignancy patients who are receiving anti-cancer treatments, such as radiation therapy and/or chemotherapy.
6. Patients with severe and/or uncontrolled medical conditions,
7. Patients on chronic corticosteroid therapy
8. A history of HIV seropositivity
9. Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study;
10. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus;
11. Uncontrolled diabetes mellitus
12. Patients who have any severe and/or uncontrolled medical conditions
13. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus;

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orrin Devinsky, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Leitner DF, Kanshin E, Askenazi M, Siu Y, Friedman D, Devore S, Jones D, Ueberheide B, Wisniewski T, Devinsky O. Pilot study evaluating everolimus molecular mechanisms in tuberous sclerosis complex and focal cortical dysplasia. PLoS One. 2022 May 19;17(5):e0268597. doi: 10.1371/journal.pone.0268597. eCollection 2022. PMID 35587487

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Subjects: This group will be treated with everolimus 7-28 days prior to surgery Everolimus: This study will measure if the drug called Everolimus effects mTOR signaling (an electrical activity signal in the brain) in patients with Tuberous Sclerosis Complex (TSC) and Focal Cortical Dysplasia (FCD) with treatment resistant epilepsy (TRE) who will be undergoing brain surgery. One group of patients will be treated with Everolimus, for 7-28 days prior to epilepsy surgery and another will not. We will determine if there is a difference in mTOR signaling between the patients who were treated with Everolimus and those who were not
Period: Overall Study
Arm/Group | Treated Subjects | Reference Subjects
Started | 5 | 10
Completed | 4 | 10
Not Completed | 1 | 0
Not completed — Surgery postponed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treated Subjects | Reference Subjects | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.25 (10.1) | 13.1 (12.3) | 14.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: .Adverse event monitoring should be continued for at least 30 days (or 5 half-lives, whichever is longer) following the last dose of study treatment
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Subjects | Reference Subjects
Number analyzed (Participants) | 4 | 10
Participants | 0 | 0

2. Secondary Outcome: Blood Everolimus Levels
Description: mTOR signaling in blood
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Treated Subjects | Reference Subjects
Number analyzed (Participants) | 4 | 10
ng/ml | 12.35 (5.36) | 2 (0)

3. Secondary Outcome: Blood Total VEGF Levels (Not Only VEGF-D)
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Treated Subjects | Reference Subjects
Number analyzed (Participants) | 4 | 10
pg/ml | 56.5 (46.9) | 50.85 (54.1)

4. Secondary Outcome: mTOR Brain Tissue-S6 Phosphate by Western Blot
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: normalized val-protein relative to actin
Arm/Group | Treated Subjects | Reference Subjects
Number analyzed (Participants) | 4 | 10
normalized val-protein relative to actin | 0.49 (0.54) | 0.81 (0.22)

5. Secondary Outcome: HMGB1 Expression in Brain Tissue
Description: HMGB1 expression is measured through label-free quantification (LFQ). LFQ is a method in mass spectroscopy that determines the relative amount of proteins in biological samples. The unit of measure is LFQ intensity; a higher LFQ intensity indicates greater HMGB1 expression.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: LFQ intensity
Arm/Group | Treated Subjects | Reference Subjects
Number analyzed (Participants) | 4 | 10
LFQ intensity | 14.85 (0.6) | 15.06 (0.35)

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Treated Subject: This group will be treated with everolimus 7-28 days prior to surgery
  Everolimus: This study will measure if the drug called Everolimus effects mTOR signaling (an electrical activity signal in the brain) in patients with Tuberous Sclerosis Complex (TSC) and Focal Cortical Dysplasia (FCD) with treatment resistant epilepsy (TRE) who will be undergoing brain surgery. One group of patients will be treated with Everolimus, for 7-28 days prior to epilepsy surgery and another will not. We will determine if there is a difference in mTOR signaling between the patients who were treated with Everolimus and those who were not
- Reference Subject: This group will be enrolled as reference subjects, and will be undergoing routine surgery as part of standard of care treatment. No intervention will be provided to these subjects as part of the study.
Arm/Group | Treated Subject | Reference Subject
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 0/4 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT02451696/Prot_SAP_000.pdf